CLINICAL TRIAL: NCT01719926
Title: Phase I Study Evaluating Indomethacin in Combination With Platinum-based Chemotherapy
Brief Title: Phase I Platinum Based Chemotherapy Plus Indomethacin
Acronym: PIFA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr. F.Y.F.L. de Vos, MD/PhD, UMC Utrecht
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL40487.041.12
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms
Keywords: Colorectal; Esophageal; Indomethacin; PIFA
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms | interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capecitabine/Oxaliplatin (Experimental): Patients receiving Capecitabine/Oxaliplatin chemotherapy
  Interventions: Drug: Indomethacin
- Cisplatin + Xeloda(Capecitabine) or Gemcitabine (Experimental): Patients receiving Cisplatin regimen
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Indomethacin — 3 times per day from 2 days before until 5 days after chemotherapy. Escalating dosage each cohort.

SUMMARY:
Mesenchymal stem cells (MSCs) are present in the circulation of cancer patients, and are recruited to the stroma of both the primary tumor and metastasis. Recent preclinical research has shown that in response to platinum-based chemotherapy, MSCs secrete two specific platinum-induced fatty acids (PIFAs) which induce resistance to a broad spectrum of chemotherapies. The secreted PIFAs are the fatty acid oxo-heptadecatetraenoic acid (KHT) and the omega-3 fatty acid hexadecatetraenoic acid (16:4). These PIFAs are produced via the COX-1 pathway. COX inhibitors, including indomethacin. This phase 1 study explores the safety of combining indomethacin with platinum containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histological proven malignancy receiving cisplatin combined with gemcitabine or 5FU/capecitabine. (cisplatin dose range 60-80 mg/m2) (Arm I) or CAPOX (oxaliplatin, capecitabine) (Arm II) in a 21 day cycle.
* Age ≥ 18 years
* Platinum-based chemotherapy naïve for at least 6 months.
* Subjects with at least one evaluable lesion.
* WHO Performance Status of 0 or 1.
* Female participants should be of non-child bearing potential either physiologic or by using adequate contraception, have a negative serum pregnancy test, and refrain from breast feeding.
* Written informed consent.

Exclusion Criteria:

* Known or suspected allergy or hypersensitivity to indomethacin or any agent given in association with this trial, in particular subjects who have a history of severe hypersensitivity reactions to anti-emetics (5-HT3 antagonists, metoclopramide or corticosteroids) and acetylsalicylic acid or other prostaglandin synthetase inhibitors.
* Symptomatic brain or meningeal tumors
* Subjects with seizure disorder requiring medication (such as corticosteroids or anti-epileptics).
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:
* Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
* Unstable angina pectoris
* Symptomatic congestive heart failure NYHA class ≥ 3 (see appendix 13.6)
* Myocardial infarction ≤ 6 months prior to randomization
* Serious uncontrolled cardiac arrhythmia
* Active peptic ulcer disease, gastritis, inflammatory bowel disease.
* History of active gastrointestinal bleeding
* History of cerebrovascular disease
* Bleeding diathesis
* Chronic renal disease defined as GFR (MDRD) <60 ml/min
* Absolute Neutrophil Count (ANC) < 1.5 x 109/L (< 1500/mm3)
* Platelets (PLT) < 100 x 109/L (< 100,000/mm3)
* Hemoglobin (Hgb) < 6.0 mmol/l (patients may be transfused to achieve adequate Hb)
* Partial thromboplastin time (PTT) > 1,5 x ULN
* Serum bilirubin > 1.5 ULN
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) > 3.0 x ULN (> 5 x ULN if liver metastases present)
* Patients who are unable or unwilling to comply with the protocol
* Chronic treatment with a corticosteroid agent (nebulized corticosteroids are allowed)
* Patients who received radiation therapy within 4 weeks of the start of the study
* Patients who received an experimental agent less than 4 weeks before start of the study.
* Patients who used Omega-3/omega-6 containing products, including fish oil products less than 2 weeks before start of the study.
* Chronic use of NSAID's and/or acetylsalicylic acid and/or other prostaglandin synthetase inhibitors.
* Use of anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of dose limiting toxicities at each dosage cohort | From first dose of indomethacin until 28 days after last dose of indomethacin

SECONDARY OUTCOMES:
Pharmacodynamics | During first 2 cycles of 3 weeks each
  Serum levels of mesenchymal stem cells and platinum induced fatty acids at T = pre-chemotherapy, one, two and four hours expressed in pmol/L.
Efficacy | From baseline to date of progressive disease according RECIST 1.1, approximately 9 to 18 weeks
  Efficacy will be assessed according RECIST 1.1 criteria. Progression free survival is defined as time from baseline CT scan to progressive disease according RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: F.Y.F.L. de Vos, MD/PhD, Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (3):
  - Meander Medisch Centrum, Amersfoort, Utrecht
  - the Netherlands Cancer Institute, Amsterdam
  - UMC Utrecht, Utrecht
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland